CLINICAL TRIAL: NCT05146180
Title: Interest of Parametric Positron Emission Computed Tomography Imaging in the Diagnosis of Infections on Cardiac Valve Prosthesis : PARAVA Study
Brief Title: Interest of Parametric Positron Emission Imaging in the Diagnosis of Infections on Cardiac Valve Prosthesis
Acronym: PARAVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHB18.10
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parametric positron emission computed tomography (Experimental)
  Interventions: Device: Parametric positron emission computed tomography

INTERVENTIONS:
Device: Parametric positron emission computed tomography — Patients will undergo parametric positron emission computed tomography in 15 days after the labeled polynuclear scintigraphy

SUMMARY:
The objective of this study is to determine if early parametric positron emission computed tomography is useful to diagnose cardiac prosthetic valve infections.

DETAILED DESCRIPTION:
In addition to routine examinations (biological and microbiological tests, transesophageal or transthoracic ultrasound, transesophageal or transthoracic ultrasound, and leukocyte scintigraphy) of a parametric acquisition during the positron emission computed tomography parametric acquisition during positron emission computed tomography , this examination being itself planned in a standard way.

The definitive diagnosis according to the Duke-Li criteria will be established three months later in a multidisciplinary consultation meeting.

The final diagnosis according to the Duke-Li criteria will be made three months later in a multidisciplinary consultation meeting, blinded to the results of the parametric positron emission computed tomography, and with knowledge of the results of the standard positron emission computed tomography and the entire work-up.

Results and all the complementary work-up.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to18 years,
* Effective contraception for women of childbearing age or negative pregnancy test on the day of the exam
* Good general condition. WHO ≤ 1
* Suspicion of endocarditis on a prosthetic heart valve implanted more than 3 months ago
* Labeled polynuclear scintigraphy performed within a maximum of 15 days before positron emission computed tomography
* Standard positron emission computed tomography planned as part of the extension assessment
* Informed and signed consent before any specific study procedure.
* Patient affiliated to the social security system

Exclusion Criteria:

* Presence of an active cancer in the previous three years
* Pregnancy or breastfeeding
* Poorly controlled diabetic patients
* Protected adults (under guardians or curators)
* Impossible decubitus (orthopnea, ...),
* Hypersensitivity to FDG or to one of the excipients of the radiopharmaceutical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Determination of diagnostic value of parametric positron emission computed tomography | 3 months
  area under the curve of the Ki parameter (and the Vd parameter) as a function of the presence of endocarditis diagnosed during the multidisciplinary consultation meeting at 3 months

SECONDARY OUTCOMES:
Correlation between parametric positron emission computed tomography and scintigraphy with labelled leukocytes | 3 months
  comparison between diagnosis established by parametric positron emission computed tomography and scintigraphy with labelled leukocytes

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Chastan, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No